CLINICAL TRIAL: NCT05906186
Title: Study Intestinal Complaints During Chemotherapy.
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Spaarne Gasthuis (Other)
Responsible Party: Sponsor
Other Study IDs: 2023.0026
Record Dates: First submitted 2023-06-07; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Constipation
Keywords: Kiwifruit; Chemotherapy
MeSH Terms: conditions — Constipation | interventions — alcohol acyltransferase, Actinidia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-test: Standard care: all patients who are starting their first (neo adjuvant or adjuvant) treatment with chemotherapy visit the nurse practitioner. Site effects like constipation will be discussed and the prescription of laxatives is standard care. Participants will keep a stool pattern diary during two months using the Bristol Stool Scale (BSS). During follow up the occurrence of side effect, such as nausea, diarrhea and constipation is assessed.
- Post-test: After the first four months (pre-test phase) of the study, nurse practitioners are asked, as lifestyle advice, to eat two kiwis per day instead of two pieces of fruit. A similar group of patients undergoing their first (neo-adjuvant or adjuvant) chemotherapy treatment are approached with a request to participate in the study. Participants keep a diary of defecation patterns for two months using the Bristol Stool Scale (BSS). During follow-up, the occurrence of side effects such as nausea, diarrhea and constipation will be assessed.
  Interventions: Behavioral: kiwifruit

INTERVENTIONS:
Behavioral: kiwifruit — eating two kiwifruits a day
  Groups: Post-test

SUMMARY:
Study intestinal complaints during chemotherapy. A prospective study into intestinal complaints in patients undergoing chemotherapy treatment. A pre and post implementation design is used to establish if eating two kiwi fruits per day can prevent constipation.

DETAILED DESCRIPTION:
The Medical Research Involving Human Subjects Act (WMO) does not apply to this research. Nonetheless it will be conducted according to the principals of Good Clinical Practice (GCP), privacy legislation (AVG) and Medical Treatment Agreement Act (WGBO). The consumption of eating two kiwi's a day can be seen as a slight variation on standard advice with regards to a healthy diet. Maintaining a diary may take some time from the participant but at the same time is of use during follow up visits where side effects, including the occurrence of constipation are discussed. The The study is approved by the Advisory Committee on Local Feasibility (ACLU) of the Spaarne Gasthuis.

ELIGIBILITY:
Inclusion Criteria:

1. First chemotherapy/cytostatics treatment
2. Neo-adjuvant or adjuvant treatment
3. Performance status World Health Organization (WHO) 0-1
4. Age 18+
5. Written informed consent
6. Command of the Dutch language

Exclusion Criteria:

1. Kiwi allergy
2. Patients using standard laxatives prior to the first chemotherapy/cytostatic treatment.
3. Patients with a history of bowel resection
4. Patients with stoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For this study adult patients undergoing their first neo adjuvant or adjuvant chemotherapy are included.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-30 (Estimated)

PRIMARY OUTCOMES:
1. How common are constipation symptoms in patients undergoing chemotherapy treatment? | 1 year

SECONDARY OUTCOMES:
2. Does the use of laxatives decrease when consuming two kiwi's a day? | 1 year
3. Which interventions against constipation do patients experience as the most comfortable? | 1 year

IPD SHARING:
Plan to Share IPD: No